CLINICAL TRIAL: NCT03701906
Title: Effect of a Mixture of New Probiotic Strains in the Colonization of the Gastrointestinal Tract of Preterm Infants.
Brief Title: Effect of a Mixture of New Probiotic Strains in Preterm Infants
Acronym: PREBIOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PRE/18.02
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: This is an interventional, randomized, double-blind, placebo-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus PS11603 & Bifidobacterium PS10402 (Active Comparator): A mixture of 1*10E9 colony forming unit (CFU) of Lactobacillus PS11603 and 1*10E8 CFU of Bifidobacterium PS10402 in 1 vial will be dissolved and enterally administered daily until discharge from the Neonatal Unit or until the 36th post-gestational week of age.
  Interventions: Dietary Supplement: Lactobacillus PS11603 & Bifidobacterium PS10402
- Placebo (Active Comparator): 1 vial of Placebo will be dissolved and enterally administered daily until discharge from the Neonatal Unit or until the 36th post-gestational week of age.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus PS11603 & Bifidobacterium PS10402 — Approximately 8 weeks intervention study: Participants with 0-5 days of age will start a period of 8 weeks of intervention. During this time the participants will intake one daily dose of the product that contains 1*10E9 CFU of L.salivarius PS11603 and 1*10E8 CFU of B.longum PS10402.
  Other Names: Lactobacillus PS11603 & Bifidobacterium PS10402 during 8 weeks
  Arms: Lactobacillus PS11603 & Bifidobacterium PS10402
Dietary Supplement: Placebo — 8 weeks intervention study: A 8 weeks intervention period. During the 8 weeks of intervention the participants will intake one daily dose of placebo supplement.
  Arms: Placebo

SUMMARY:
An interventional, randomized, double-blind, placebo-controlled study will be conducted to investigate the effect of a new probiotic strain Lactobacillus PS11603 & Bifidobacterium PS10402 in premature infants from 28 weeks + 0 days to 30 weeks + 6 days of gestation.

The study duration will be 2 months, which includes 8 weeks product administration. Participants will be randomized assigned to one of the two study groups: the control group with placebo consumption and a probiotic consumption group.

DETAILED DESCRIPTION:
An interventional, randomized, double-blind, placebo-controlled study will be conducted to investigate the effect of a new probiotic strains Lactobacillus PS11603 & Bifidobacterium PS10402 in 30 premature infants born within 28 weeks + 0 days to 30 weeks + 6 days of gestation.

The duration of participation in the study is estimated to be 40-60 days. Participants will be randomized assigned to one of the two arms of the study: the control group, with placebo consumption, and a probiotic consumption group. The aim of the study will be investigate the effect of the probiotics strains in the colonization of the intestinal tract of preterm babies.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between week 28 + 0 days and week 30 + 6 days of gestation.
* Written informed consent signed by the parent or legal guardian.
* Tolerate enteral feeding, at least 10mL / kg / day.
* Postnatal age ≤ 5 days

Exclusion Criteria:

* Child with malformations
* With short bowel syndrome or any surgery in the gastrointestinal tract
* With defect in the intestinal epithelial barrier

Ages: 1 Minute to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Counts (CFU/g) of Bifidobacterium and Lactobacillus colonies from fecal samples. | 2 months
  Counts (CFU/g) of Bifidobacterium and Lactobacillus presents in fecal samples from preterm infants

CONTACTS AND LOCATIONS:
Overall Officials: Susana Manzano, PhD, Study Chair — ProbiSearch SL
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moreno-Sanz B, Montes MT, Manzano S, Espinosa-Martos I, Cardenas N, Esteban S, Cruz M, Jimenez E, de Pipaon MS. Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effect of Two Probiotics on the Preterms' Gut Microbiota. J Pediatr Gastroenterol Nutr. 2022 Jun 1;74(6):e153-e159. doi: 10.1097/MPG.0000000000003427. Epub 2022 Feb 25. PMID 35221319